CLINICAL TRIAL: NCT05693545
Title: Intramuscular vs. Enteral Penicillin Prophylaxis to Prevent Progression of Latent Rheumatic Heart Disease: A Non-inferiority Randomized Trial
Brief Title: GOALIE: Intramuscular vs. Enteral Penicillin Prophylaxis to Prevent Progression of Latent RHD Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0892
Record Dates: First submitted 2023-01-04; First posted 2023-01-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Penicillin V; Penicillin G

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Pencillin (Experimental): Oral phenoxymethyl penicillin (Pen V) prophylaxis 250mg twice daily.
  Interventions: Drug: phenoxymethyl penicillin
- IM Penicillin (Active Comparator): Intramuscular benzathine benzylpenicillin G (BPG) prophylaxis (600,000 IU for children <30kg, 1.2 million IU for children ≥30kg), every 28 days
  Interventions: Drug: intramuscular benzathine penicillin G (BPG) prophylaxis

INTERVENTIONS:
Drug: phenoxymethyl penicillin — Prophylaxis
  Other Names: Pen V
  Arms: Oral Pencillin
Drug: intramuscular benzathine penicillin G (BPG) prophylaxis — Prophylaxis
  Other Names: benzathine penicillin G, BPG, penicillin prophylaxis
  Arms: IM Penicillin

SUMMARY:
The goal of this clinical trial is to determine if twice daily oral penicillin prophylaxis is non-inferior to monthly IM penicillin prophylaxis in preventing latent Rheumatic Heart Disease Progression in children between the ages of 5-17 years. The main objective is to compare the proportion of children aged 5-17 years with latent RHD receiving oral penicillin prophylaxis who progress to worse valvular disease at 2-years compared to children who receive IM penicillin prophylaxis.

DETAILED DESCRIPTION:
GOALIS is a randomized controlled trial developed to provide high quality contemporary evidence on the efficacy of oral penicillin as RHD prophylaxis.

Aim 1: To compare the proportion of children aged 5-17 years with latent RHD receiving oral penicillin prophylaxis who progress to worse valvular disease at 2-years compared to children who receive IM penicillin prophylaxis.

Aim 2: To evaluate the economic equivalence and cost-effectiveness of oral penicillin compared to IM penicillin, after echocardiographic screening for latent RHD detection.

Aim 3: Compare patient-reported outcomes (treatment acceptance, treatment satisfaction, and health-related quality of life) between children receiving oral and IM penicillin prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Has a new diagnosis of latent RHD detected through primary or secondary school echocardiographic screening.
* Has agreed to participate in the study via the study's informed consent/assent process.

Operational Definition of Latent RHD Borderline RHD or Mild Definite RHD (to include no more than mild regurgitation at the mitral or aortic valve, normal mean mitral and aortic valve gradients, normal bi-ventricular function) according to the 2012 WHF consensus criteria.

Exclusion Criteria:

* Known history of ARF or RHD
* Newly diagnosed RHD by echo screening considered to be "missed clinical RHD" as compared to true latent RHD including: > mild pathological valvular regurgitation at the mitral valve or aortic valve, mitral stenosis (mean MV gradient ≥ 4mmHg) (definite B61), aortic stenosis (mean AV gradient ≥ 20mmHg)
* Structural or functional cardiac defects, other than those consistent with RHD, that were known prior to or detected through echo screening (except patent foramen ovale, small atrial septal defect, small ventricular septal defect, small patent ductus arteriosus)
* Self-report of prior allergic reaction to penicillin
* Any known conditions predisposing to thrombocytopenia or hypercoagulability, or other contraindications to intramuscular injection
* Any known co-morbid conditions (ex. HIV, renal deficiencies, severe malnutrition) that have resulted in prescription of regular antibiotic prophylaxis)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1004 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression | 2 year endpoint
  Progression of echocardiographic features of latent RHD to borderline to definite, or definite to mild or definite to moderate/severe

SECONDARY OUTCOMES:
Demonstrate non-inferior costs and cost-effectiveness of oral penicillin compared to IM penicillin | baseline, 6, 12, 18, 24 months post randomization
  The aim is to understand the costs and effectiveness of the intervention. Costs will include intervention and disease specific costs, capturing both health system and family out of pocket costs. Participants will complete a questionnaire asking about out-of-pocket cost (medications, supplies, consultation fees) and lost productivity (including missed school and workdays) due to the intervention. Costs will be measured in the local currency (Uganda Shillings) and presented in United States dollars (USD)
Obtain cost data associated with the receipt of oral or IM penicillin in the community from a healthcare provider perspective. | 2 year endpoint
  In order to understand health center and community costs, 10 randomly selected health care facilities (including level II, III, and IV facilities) will be surveyed to obtain direct costs of medications, supplies as well as any administration and professional fees associated with outpatient and inpatient visits.
Treatment Acceptance | baseline, 6, 12, 18, 24 months post randomization
  Treatment acceptance will be assessed with the widely-used Chronic Treatment Acceptance (ACCEPT) questionnaire, a generic medication acceptance instrument validated for chronic conditions. This 25-item survey consists of six areas of focus: medication convenience (3 items), length of treatment (2 items), medication constraints (9 items), medication side effects (5 items), medication effectiveness (3 items), medication advantages (3 items). Responses are rated on a 5-point Likert scale and scores of 1 through 4 indicating increasing levels of acceptance.
Treatment Satisfaction | baseline, 6, 12, 18, 24 months post randomization
  Treatment Satisfaction will be assessed with the 14-item Abbreviated Treatment Satisfaction Questionnaire (v 1.4). This widely used survey contains 4 areas of focus including satisfaction of treatment effectiveness (3 items), satisfaction with treatment side effects (5 items), satisfaction with treatment convenience (3 items), and a global treatment satisfaction (3 items). Scores are then transformed to a score of 0-100 to create the overall scale score and the subcategory scores, with higher scores representing higher treatment satisfaction on that domain.
Health-Related Quality of Life | baseline, 6, 12, 18, 24 months post randomization
  Health Related Quality of Life will be measured using the Pediatric Quality of Life Inventory Version 4.0 Generic Core (PedsQL 4.0) questionnaire. The PedsQLTM4.0 is a 23-item survey for children aged 5-18 which assesses HRQOL. It has four areas of focus: Physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), school functioning (5 items). Each item has five possible responses measuring the extent to which the item was a problem during the past month. The possible responses are measured using a 5-point Likert scale from 0=never a problem to 4 = almost always a problem. These reverse scaled scores are then transformed to a score of 0-100 to create the overall scaled score and the subcategory scores, with higher scores representing better quality of life.
Patient-reported outcomes | baseline, 6, 12, 18, 24 months post randomization
  Interviews will be used to collect qualitative data around participants perceptions of the impact of RHD and its treatment on their activities of daily living and quality of life including experiences with IM or oral penicillin prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z Beaton, Principal Investigator — Cincinnati Chidren's hospital
Locations (1):
- Uganda Heart Institute, Kampala, Uganda

REFERENCES:
- [Derived] Rwebembera J, Ndagire E, Carvalho N, Webel AR, Sable C, Okello E, Sarnacki R, Spaziani AM, Mucunguzi A, Engelman D, Grobler A, Steer A, Beaton A. Intramuscular versus enteral penicillin prophylaxis to prevent progression of rheumatic heart disease: Study protocol for a noninferiority randomized trial (the GOALIE trial). Am Heart J. 2024 Sep;275:74-85. doi: 10.1016/j.ahj.2024.05.012. Epub 2024 May 24. PMID 38797460